CLINICAL TRIAL: NCT05502328
Title: Radicle™ Energy: A Randomized, Blinded, Placebo-controlled Study of Cannabinoid Formulations and Their Effects on Energy Levels, Focus, Appetite and Other Health Outcomes
Brief Title: Radicle Energy: A Study of Cannabinoids on Energy and Other Health Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radicle Science (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: RADX-22D02
Record Dates: First submitted 2022-08-08; First posted 2022-08-16 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Energy

STUDY DESIGN:
Intervention Model Description: Participants will be stratified based on gender and endorsement of problems with energy and/or focus reported during enrollment, then randomized to one of the study arms
Who Masked: Participant, Investigator
Masking Description: The investigator is blinded to the participants assigned study products. Participants are blinded to the study product they received.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Control 1 (Placebo Comparator): Energy Product Form 1 - control
  Interventions: Dietary Supplement: Energy Study Product Usage
- Control 2 (Placebo Comparator): Energy Product Form 2 - control
  Interventions: Dietary Supplement: Energy Study Product Usage
- Energy Product 1.1 (Experimental): Energy Product Form 1 - active product 1
  Interventions: Dietary Supplement: Energy Study Product Usage
- Energy Product 1.2 (Experimental): Energy Product Form 1 - active product 2
  Interventions: Dietary Supplement: Energy Study Product Usage
- Energy Product 2.1 (Experimental): Energy Product Form 2 - active 1
  Interventions: Dietary Supplement: Energy Study Product Usage
- Energy Product 2.2 (Experimental): Energy Product Form 2 - active 2
  Interventions: Dietary Supplement: Energy Study Product Usage

INTERVENTIONS:
Dietary Supplement: Energy Study Product Usage — Participants will use their Radicle Energy study product as directed for a period of 4 weeks.

SUMMARY:
A randomized, blinded, placebo-controlled study of cannabinoid formulations and their effects on energy levels, focus, appetite and other health outcomes

DETAILED DESCRIPTION:
This is a randomized, blinded, placebo-controlled study conducted with up to 300 adult participants per study arm (3000 total), age 21 and older and residing in the United States.

Eligible participants will (1) endorse a desire for more energy (less fatigue and/or better concentration/focus during screening); (2) indicate a willingness to refrain from taking cannabinoids during the study period, and (3) indicate an interest in taking a plant derived cannabinoid product to help with their energy and/or focus.

Participants with known liver disease, heavy drinkers, and those who are pregnant, trying to become pregnant, or breastfeeding will be excluded. Those taking medications that warn against grapefruit consumption will be excluded. People with a calculated BMI of 18.5 or less will be excluded.

Self-reported data are collected electronically from eligible participants over 5 weeks. Participant reports of health indicators will be collected during baseline, throughout the active period of study product use, and in a final survey. All study assessments will be electronic; there are no in-person visits or assessments for this real-world evidence study.

ELIGIBILITY:
Inclusion Criteria:

* 21 years of age and older
* Resides in the United States
* Endorses: a desire for more energy (less fatigue) and/or a desire for better concentration (focus/attention)
* Selects more energy and/or better concentration as a primary reason for taking a cannabinoid product
* Expresses a willingness to refrain from taking any non-study cannabinoid product (i.e.

CBD, THC) for the duration of participant engagement

* Expresses a willingness to take a study product and not knowing the product identity until the end of the study

Exclusion Criteria:

Pregnant, trying to become pregnant, or breastfeeding Reports a diagnosis of liver disease Reports being a heavy drinker (defined as drinking 3 or more alcoholic beverages per day) Unable to read and understand English Lack of reliable daily access to the internet Reports taking any medication that warns against grapefruit consumption Calculated BMI 18.5 or less

Ages: 21 Years to 105 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1427 (Actual)
Dates: Start 2022-08-17 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-05-24 (Actual)

PRIMARY OUTCOMES:
Change in energy | 4 weeks
  Change in mean energy score as assessed by Patient Reported Outcome Measurement System (PROMIS) Fatigue 7a (scale 1-5; where lower score is less fatigue)
Change in focus | 4 weeks
  Change in concentration (ability to focus) score as assessed by PROMIS™ Cognition 6a (scale 1-5; where lower score is worse focus (cognitive function))

SECONDARY OUTCOMES:
Change in energy (measure 2) | 4 weeks
  Change in energy level score as assessed by a visual analog scale (VAS; Scoring from 0 to 10, with 0 being 'No energy' and 10 being 'More than enough energy')
Change in body weight | 4 weeks
  Change in body weight as assessed by self-reported body weight in pounds
Change in appetite | 4 weeks
  Change in appetite as assessed by a visual appetite scale (VAS; Scoring from 0 to 10, with 0 being 'No hunger' and 10 being 'Always hungry')
Change in overall quality of life (QOL) | 4 weeks
  Change in QOL score as assessed by Kemp QOL (scale 1-7; with higher scores corresponding to higher quality of life)
Change in overall well-being | 4 weeks
  Change in well-being score as assessed by World Health Organization 5 Well-being Index (WHO-5 Well-being Index; with higher scores corresponding to greater well-being)

OTHER OUTCOMES:
Change in pain | 4 weeks
  Change in pain score as assessed by the Pain on average, Enjoyment of life, and General activity Score (PEG; scale 0-10 where 0 is no pain)
Change in Sleep quality | 4 weeks
  Change in sleep quality (sleep disturbance) score as assessed by the PROMIS Sleep Disturbance 4A (scale 4 to 20; where higher scores correspond to higher levels of sleep disturbance)
Change in feelings of anxiety | 4 weeks
  Change in anxiety score as assessed by the PROMIS Anxiety 4a (scale 4-20; where higher scores correspond to greater levels of anxiety)
Change in Stress | 4 weeks
  Change in stress score as assessed by the PROMIS Stress 4a (scale 4-20; where higher scores correspond to greater levels of stress)

CONTACTS AND LOCATIONS:
Overall Officials: Emily K Pauli, PharmD, Principal Investigator — Radicle Science Inc.
Locations (1):
- Radicle Science, Inc, Del Mar, California, United States

IPD SHARING:
Plan to Share IPD: No
Data will not be shared with researchers outside of Radicle Collaborators on this study.

REFERENCES:
- See also: Radicle Science, Inc — http://radiclescience.com